CLINICAL TRIAL: NCT00463021
Title: A Phase 4, Multi Center, Open-Label, Randomized Study to Determine Clinically Appropriate Doses of Hectorol® (Doxercalciferol Capsules) When Converting From Zemplar® (Paricalcitol Injection) for the Treatment of Secondary Hyperparathyroidism in Stage 5 Chronic Kidney Disease (CKD) Subjects on Hemodialysis.
Brief Title: A Phase 4 Study to Determine Dosing of Hectorol® Capsules When Converting From Zemplar® Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HECT00306
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Hectorol (doxercalciferol capsules); Zemplar (paricalcitol injection)
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — 1 alpha-hydroxyergocalciferol; paricalcitol

INTERVENTIONS:
Drug: Hectorol (doxercalciferol capsules)
Drug: Zemplar (paricalcitol injection)

SUMMARY:
Protocol HECT00306 aims to determine clinically appropriate doses of Hectorol (doxercalciferol capsules) when converting from Zemplar (paricalcitol injection) for the treatment of secondary hyperparathyroidism in Stage 5 chronic kidney disease on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be receiving hemodialysis three times per week for a minimum of six months.
* The subject must have been receiving Zemplar Injection for a minimum of 3 months. The subject must have been on a stable dose regimen, three times per week administration for a minimum of four weeks.
* The central laboratory assessment must be within the following ranges: serum iPTH between 150-600 pg/mL, inclusive; corrected calcium < 10.0 mg/dL; phosphorus < 7.0 mg/dL.

Exclusion Criteria:

* In the opinion of the Investigator, the subject currently has poorly controlled diabetes mellitus, poorly controlled hypertension, active vasculitis, HIV infection, or any other clinically significant, unstable medical condition.
* Abnormal liver function as measured by ALT/AST greater than two times the upper limit of normal (ULN).
* The subject currently has malabsorption, severe chronic diarrhea, or ileostomy.
* Any evidence of active malignancy except for basal cell carcinoma of the skin. A history of malignancy is not an exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-04; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Dose Conversion | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- United States (8):
  - Downey, California
  - Paramount, California
  - Hudson, Florida
  - Augusta, Georgia
  - Decatur, Georgia
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Norfolk, Virginia

REFERENCES:
- See also: US FDA Approved Full Prescribing Information for Hectorol® Capsules — http://www.hectorol.com/docs/Hectorol%20Capsule%20PI%20Text_2006-01.pdf